CLINICAL TRIAL: NCT06258863
Title: Investigating the Effects of Different Incision Types on Aesthetic Outcomes and Incision-related Complications After Breast Reconstruction Surgery
Status: Enrolling by invitation | Type: Observational
Sponsor: Hubei Cancer Hospital (Other)
Responsible Party: Principal Investigator, Xinhong Wu, PhD, Chief Physician, Hubei Cancer Hospital
Other Study IDs: LLHBCH2023YN-046
Record Dates: First submitted 2024-01-15; First posted 2024-02-14 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-11

CONDITIONS: Breast Neoplasm Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- inframammary fold incision: A total mastectomy was performed using an inframammary fold incision
  Interventions: Procedure: incision type
- lateral chest wall incision: A longitudinal incision was made in the lateral chest wall for a total mastectomy
  Interventions: Procedure: incision type
- circumareolar incision: A total mastectomy was performed with an arc-shaped incision around the areola without limiting the distance to the nipple
  Interventions: Procedure: incision type
- radial incision: A total mastectomy was performed with a radial incision around the nipple
  Interventions: Procedure: incision type

INTERVENTIONS:
Procedure: incision type — Total mastectomy was performed using one of the four incision types

SUMMARY:
1. DATA COLLECTION: About 300 cases of female patients who underwent breast reconstruction at Hubei Cancer Hospital(HBCH) between February 2013 and June 2023 were retrospectively collected. The incision was defined as the mastectomy incision and was grouped by the commonly used inframammary fold incision, lateral chest wall incision, circumareolar incision, and radial incision. The incidence of postoperative incision-related complications was recorded for different incision types;
2. DATA ORGANIZATION: Patients were divided into subgroups based on history of previous breast surgery, location and size of the lump, retention of the nipple-areola complex, timing of reconstruction, and type of the implant. The correlation of each subgroup with incision design is discussed;
3. FOLLOW-UP: Collected cases were followed up by telephone to complete the Breast-Q questionnaire (aesthetic score);
4. DATA ANALYSIS: The incidence of postoperative incision-related complications and aesthetic scores for different incision types were statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. total mastectomy
2. implant and/or autologous breast reconstruction.

Exclusion Criteria:

1. No total mastectomy
2. loss of data or loss of follow-up
3. fatal cases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: About 300 female patients who underwent breast reconstruction at Hubei Cancer Hospital between January 2019 and September 2023 were collected.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2025-11-18 (Estimated)

PRIMARY OUTCOMES:
Breast-Q Version 2.0 Reconstruction Module | three months after surgery; six months after surgery; 1 year after surgery
  The questionnaire was filled in by the subjects, and the researchers assigned scores according to the results of the questionnaire. scores of the following three parts were recorded according to the Breast-Q Version 2.0© reconstruction module, with higher scores indicating better aesthetic results, Psychosocial Well-being (0 to 100), Sexual Well-being (0 to 100), Satisfaction with Breasts (0 to 100)

SECONDARY OUTCOMES:
Incision-Related Complications | within 1 year after surgery
  The researchers followed up the patients closely after surgery, and recorded the incidence of different postoperative incision complications of the subjects, such as infection, seroma, incision dehiscence, and capsular contracture.

CONTACTS AND LOCATIONS:
Locations (1):
- Hubei Cancer Hospital, Wuhan, Hongshan District, China